CLINICAL TRIAL: NCT06967987
Title: Open-label Non-randomized Multicentric Phase 2 Study Evaluating the Combination of Bemarituzumab + FLOT Chemotherapy in Perioperative Setting for Resectable Stage cT2-T4a or N+ Gastric and GEJ Adenocarcinoma Overexpressing FGFR2b
Brief Title: Study Evaluating the Combination of Bemarituzumab + FLOT Chemotherapy in Perioperative Setting for Resectable Stage cT2-T4a or N+ Gastric and GEJ Adenocarcinoma Overexpressing FGFR2b
Acronym: BEMAFLOT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation of product manufacturing by the funder prior to the start of participant enrollment
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Amgen Ltd., United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2023-10; 2024-514078-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gastric and Gastro-oesophageal Junction (GEJ) Adenocarcinomas; Overexpression FGFR2b
Keywords: Gastric and gastro-oesophageal junction (GEJ) adenocarcinomas; Resectable non-metastatic cT2-T4NX; FLOT regimen; Bemarituzumab
MeSH Terms: conditions — Adenocarcinoma | interventions — bemarituzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bemarituzumab + Flot regimen (Experimental)
  Interventions: Drug: Bemarituzumab + Flot regimen

INTERVENTIONS:
Drug: Bemarituzumab + Flot regimen — Bemarituzumab (IV administration) over 30 min (+/- 10min) at C1D1 to C8D1 + 15 mg/kg of bodyweight + single additional dose of 7,5 mg/kg at C1D8
  + FLOT regimen
  * Fluorouracil for solution for infusion (IV administration) as a continuous IV infusion approximately 24 hours 2600 mg/m²
  * Leucovorin (folinic acid) solution for infusion (IV administration) over 120 min on the first day, 200 mg/m²
  * Oxaliplatin concentrate for solution for infusion (IV administration) over 120 min on the first day, 85 mg/m²
  * Docetaxel concentrated for solution for infusion (IV administration) over 60 min on the first day, 50 mg/m²

SUMMARY:
Gastric and gastro-oesophageal junction (GEJ) adenocarcinomas rank as the fifth leading cause of cancer globally. The standard treatment for resectable non-metastatic cT2-T4NX gastric or GEJ adenocarcinoma is perioperative FLOT chemotherapy. In the FLOT4 trial, which included 55% of GEJ and 45% of gastric tumours, the FLOT chemotherapy regimen improved both disease-free survival and overall survival compared to the ECF/ECX regimen. The median overall survival was 50 months, and median disease-free survival was 30 months for the FLOT experimental arm. About 16% of patients achieved a pathological complete regression (TRG1a) in the modified ITT population treated by FLOT. For GEJ adenocarcinoma, the ESOPEC trial has recently demonstrated the superiority of FLOT regimen compared to radiochemotherapy (CROSS regimen) [ median overall survival 66 months for FLOT regimen vs 37months [HR 0.7 95% IC (0.53-0.92) p= 0.012].

Genomic analyses of gastric and GEJ adenocarcinomas conducted by the Cancer Genome Network Atlas have identified four distinct subtypes of tumours based on their gene expression profile. These subtypes include tumours positive for Epstein-Barr virus, microsatellite unstable tumours, genomically stable tumours, and tumours with chromosomal instability. This research has identified oncogenic driver alterations, leading to new targeted therapies and therapeutic strategies.

HER2 amplification and MSI status are current targets for targeted therapies with anti-HER2 antibodies and Immune Checkpoint Inhibitors (ICI), respectively. Trials using these therapies in perioperative settings are ongoing with promising preliminary results. However, targeted therapies are not currently available in the non-metastatic setting.

The overexpression of Fibroblast Growth Factor Receptor 2 (FGFR2) is a frequent molecular alteration in gastric and GEJ tumours, presenting a potential new therapeutic target. FGFR2b overexpression is associated with poor prognosis and can be detected through pre-screening by immunohistochemistry. Bemarituzumab, a monoclonal antibody specific to the splice-variant FGFR2b, has shown promising results in combination with chemotherapy in phase 2 trials.

Based on the frequency of FGFR2b overexpression, the tolerability of combination therapy with chemotherapy, and the need to improve survival rates for gastric and GEJ cancer patients, it is proposed to test the efficacy of the combination of FLOT chemotherapy and bemarituzumab in the perioperative setting for c T2-T4a or N+ gastric or GEJ adenocarcinoma MSS and overexpressing FGFR2b.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed and dated an informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol. A signed informed consent must be obtained prior to conducting any study-specific procedures
* Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Participants must have histologically confirmed diagnosis of gastric or gastroesophageal junction (Siewert 2-3) adenocarcinoma
* Tumour archival tissue must be provided for analysis of FGFR2b overexpression prior to inclusion
* Positive FGFR2b overexpression status by immunohistochemistry was defined as exhibiting any moderate (2+) to strong (3+) membranous staining in ≥ 10% of tumour cells.
* ECOG performance status score of 0 or 1
* cT2-T4a or N+ made by CT scan and endoscopic ultrasound and according to UICC 8e edition gastric or gastroesophageal junction (Siewert 2-3) adenocarcinoma without distant metastases (M0), without infiltration of adjacent structures or organs. If peritoneal carcinomatosis is clinically suspected, laparoscopic exclusion of peritoneal carcinomatosis is mandatory
* Adequate hematologic and organ function as assessed by the following laboratory tests performed within 7 days before start of study treatment:
* Male and female adult participants 18 years of age or more
* Affiliated to French social regimen
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception during treatment and for an additional 90 days after the last dose of bemarituzumab, 15 months after the end of the treatment with oxaliplatin, 6 months after the end of the treatment with fluorouracil, 2 months after the end of the treatment with docetaxel
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study intervention during treatment and for an additional 6 months after the last dose of bemarituzumab, 12 months after the end of the treatment with oxaliplatin, 3 months after the end of the treatment with fluorouracil and 4 months after the end of the treatment with docetaxel

Exclusion Criteria:

* Distant metastases or infiltration of adjacent structures or organs and all primarily non-resectable stages. Patients with enlarged, metastasis suspected, para-aortal, mesenterial or para pancreatic lymph nodes are M1 and must not be enrolled into the trial
* Loss of body weight ≥10% in the month before inclusion
* Other histology than adenocarcinoma.
* Tumour with microsatellite instable disease detected by ICH or NGS are excluded
* History of peripheral neuropathy with symptoms≥ grade 2
* Known allergy, hypersensitivity or contraindication to components of bemarituzumab formulation including polysorbate
* History of systemic disease or ophthalmologic disorders requiring chronic use of ophthalmic steroids
* Ocular related disorders:
* History of systemic disease or ophthalmologic disorders requiring chronic use of ophthalmic steroids
* Evidence of any ongoing ophthalmologic abnormalities or symptoms that are acute (within 4 weeks) or are actively progressing
* Recent (within 6 months) corneal surgery or ophthalmic laser treatment or recent (within 6 months) history of, or evidence of, corneal defects, corneal ulcerations, keratitis, or keratoconus, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer
* Unwillingness to avoid use of contact lenses during study treatment and for ≥ 100 days after the end of treatment
* Prior immunosuppressive therapy: immunosuppressive doses of systemic medications of > 10 mg/day of prednisone or equivalent must be discontinued ≥ 2 weeks before the first dose of study treatment. Short courses of high dose corticosteroids and/or continuous low dose of prednisone (< 10 mg/day) are permitted. In addition, inhaled, intranasal, and/or joint injections of corticosteroids are allowed.
* Chronic inflammatory intestinal disease
* Known allergy, hypersensitivity or contraindication against 5-Fluorouracil, Leucovorin, Oxaliplatin, Docetaxel or Bemarituzumab
* Severe acute disease or active infection requiring systemic treatment or any uncontrolled infection within 14 days before the first dose of study treatment
* History of cardiac disorders as defined by: Congestive heart failure ≥ New York Heart Association (NYHA) class 2, acute myocardial infarction < 6 months prior or evolutive cardiopathy to the first dose of study treatment, unstable angina within 6 months before the first dose of study treatment, acute myocardial infarction < 6 months prior to the first dose of study treatment, uncontrolled hypertension (defined as an average systolic blood pressure >160 150 mmHg or diastolic >100 90 mm Hg despite optimal treatment (measured following European Society for Hypertension/European Society of Cardiology [ESH/ESC] 2018 guidelines); uncontrolled cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, active coronary artery disease, QTc ≥ 470ms
* No reversible electrolyte disorders such as hypokalemia, hypocalcemia or hypomagnesemia
* Any haemorrhage or bleeding event ≥ NCI-CTCAE Grade 3 within 28 days prior to the start of study treatment
* Known human immunodeficiency virus infection with CD4+ T cell counts < 350 cells/µL, hepatitis C infection (subjects with hepatitis C who achieve a sustained virologic response following antiviral therapy are permitted), or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody who achieve sustained virologic response with antiviral therapy directed at hepatitis B are permitted)
* Subjects who experienced severe, life-threatening, or recurrent (Grade 2 or higher) immune-mediated adverse events (AEs) or infusion-related reactions including those that led to permanent discontinuation while on treatment with immune-oncology agents
* History of other malignancy within the past 2 years with exception of skin non melanoma cancer and in situ carcinoma of cervix
* Major contra indication to surgery including cirrhosis, oesophageal varices, severe respiratory insufficiency VEMS <1L and severe obliterating arteriopathy of the lower limbs.
* Partial or total DPD deficiency
* History or evidence of any other clinically significant disorders, conditions, or diseases that in the opinion of the investigator or sponsor, if consulted, would pose a risk to subject safety, or interfere with study procedures or completion
* Participation in another therapeutic clinical study or receiving any investigational agent within 28 days of enrolment or during this clinical study
* Live attenuated vaccines
* Recent (in the last 4 weeks) or concomitant treatment with brivudine.
* Female subjects of childbearing potential unwilling to use highly effective methods of contraception during treatment and for an additional 90 days after the last dose of bemarituzumab, 15 months after the end of the treatment with oxaliplatin, - 6 months after the end of the treatment with fluorouracil - 2 months after the end of the treatment with docetaxel
* Female subjects who are breastfeeding or who plan to breastfeed while on the study through 90 days after the last dose of bemarituzumab
* Female subjects planning to conceive while on the study through 90 days after the last dose of bemarituzumab
* Male who are sexually active with WOCBP unwilling to use highly effective methods of contraception during treatment and for an additional 90 days after the last dose of bemarituzumab during treatment, 12 months after the end of the treatment with oxaliplatin,3 months after the end of the treatment with fluorouracil, 4 months after the end of the treatment with docetaxel
* Female subjects of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive serum pregnancy test
* Subject likely to be unavailable to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the efficacy of a combination of FLOT chemotherapy with bemarituzumab as perioperative treatment for gastric and GEJ adenocarcinoma. | 6 months
  The primary endpoint is the complete pathological response in histological result of primary tumour and lymph nodes from the surgical resection, using Becker tumour scale (TG1 to TG3) from TG1 (a and b) to TG2 resection grading

CONTACTS AND LOCATIONS:
Overall Officials: Judith Raimbourg, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (12):
- France (12):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Bergonié, Bordeaux
  - CHRU de Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to concerns regarding participant privacy and the lack of explicit consent for data sharing beyond the scope of the current study."